CLINICAL TRIAL: NCT02376634
Title: The Effectiveness of Clinical Hypnotherapy in Reducing Anxiety and Pain in Major Surgical Procedures (Nuss and Scoliosis Repair)
Brief Title: Hypnotherapy in Major Surgical Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Nationwide Children's Hosp.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Haleh Saadat, Director of Complementary and Alternative Medicine, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB14-00837
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-07

CONDITIONS: Scoliosis; Pectus Excavatum
MeSH Terms: conditions — Scoliosis; Funnel Chest | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis (Active Comparator): The hypnosis group will receive a semi-structured intervention by primary investigator. The intervention is somewhat individualized based on the recipients personal characteristics (e.g., age, gender, medical history). The intervention will begin with an "induction" phase during which the participant is guided to relax and to focus their attention on one stimuli. The intervention will then proceed with a "suggestion" phase. Suggestions used in this phase will all be directed toward decreasing the patient's anxiety and post-operative pain. Patients will be taught self-hypnosis to decrease distress and reframe painful experiences.
  Interventions: Behavioral: Hypnosis
- Control (No Intervention): This group will receive the standard of care of Nationwide Children's Hospital.

INTERVENTIONS:
Behavioral: Hypnosis — Patients will be taught self-hypnosis.
  Arms: Hypnosis

SUMMARY:
The purpose of this randomized controlled study is to test the feasibility of clinical hypnotherapy as a perioperative intervention for the reduction of pre-operative anxiety, post-operative pain, and other-related symptoms (nausea, vomiting, spasms, length of stay, self mastery) in children undergoing scoliosis repair or Nuss procedure.

DETAILED DESCRIPTION:
Participants will be 60 children, aged 10-21, ASA 1 and 2 Classification, with idiopathic scoliosis or congenital deformity of the chest wall, who are undergoing Nuss procedure/scoliosis repair at the Nationwide Children's hospital. The design of this study is a single-blinded randomized controlled trial-comparing pre-operative anxiety, post-operative pain and other related symptoms in two groups of:

Group 1: Receives hypnosis (described below) Plus PCA Group 2: Standard of care (PCA)

Interventions:

Group I) Hypnosis: The hypnosis group will receive a semi-structured intervention by primary investigator. The intervention is somewhat individualized based on the recipients personal characteristics (e.g., age, gender, medical history). The intervention will begin with an "induction" phase during which the participant is guided to relax and to focus their attention on one stimuli. The intervention will then proceed with a "suggestion" phase. Suggestions used in this phase will all be directed toward decreasing the patient's anxiety and post-operative pain. Patients will be taught self-hypnosis to decrease distress and reframe painful experiences.

Group II) Control: This group will receive the standard of care of Nationwide Children's hospital.

Procedures:

1. Potential participants will be identified through review of the NCH surgery schedule and assessed for eligibility by review of the electronic medical record using the exclusionary criteria listed below.
2. In order to assure valid data, all anesthetic protocol will be standardized.
3. All patients will be randomized to the Hypnosis group and control group by another member of the research team based on a randomization table. The patient's group assignment will be placed in a sealed envelope prior to the day of surgery. Only PI can access the envelope prior to the intervention. The PI will only perform the assigned intervention while the research assistant and other health care providers are not present. The research assistant and the peri-operative health care personnel will remain blind to group assignment throughout data collection.
4. A research assistant will administer a brief assessment of state of anxiety (STAI) that will take the patient at most 5 minutes to complete.
5. The research assistant will measure patient's blood pressure (BP) and heart rate (HR).
6. The PI will perform the clinical hypnotherapy intervention and teach self-hypnosis at two points of time in Hypnosis group;

   1. In pre-op visit prior to the surgery date
   2. on the day of, prior to the procedure
7. A second research assistant will administer a second brief assessment of anxiety (STAI), and measure HR and BP again.
8. Once the patient enters the operating room the standardized anesthetic protocol ( as describe below) will be employed.
9. Following surgery, in the Post Anesthesia Care Unit (PACU) and floors we standardize pain management with PCA orders.
10. Postoperative analgesia will be provided by hydromorphone delivered via a patient-controlled analgesia (PCA) device with a bolus dose of 4-8 µg/kg and a lockout period of 8-10 minutes. This may be increased up to 10 µg/kg as needed to achieve optimal analgesia. No basal infusion will be administered for the PCA. The nursing staff in post-anesthesia recovery unit and study staff collecting post-operative pain scores until 24 hours post-operatively will be blinded as to the group assigned. The subject's pain scores will be collected and recorded using the Visual Analogue Scale (VAS) pain scale. Total opiate consumption in the first 24 hours will be recorded. The need for medications to treat opiate-related side effects including naloxone or ondansetron for pruritus or nausea respectively will be recorded. We will record the number of deliveries and demands from the PCA device. We will also record the length of hospital stay.

Measures

* State-Trait Anxiety Inventory (STAI)15. The STAI, completed by the patient to chart their own anxiety level, is a 40-item self-report measure that contains 20 items measuring state anxiety and 20 items measuring trait anxiety. Subjects are asked to respond on a 4-point Likert scale. Total scores for state and trait portions separately range from 20 to 80, with higher scores denoting higher levels of anxiety.
* Visual Analog Scale (VAS) The VAS is completed by the blind observer to chart their own rating of the patient's pain. It is a 10cm line where the observer can mark a line anywhere from "not anxious at all" to "very anxious"
* McGill Pain Questionnaire (MPQ). Sensory and effective dimensions of pain are measured using the short MPQ, which consists of 15 pain descriptors that are rated on a 4-point severity scale from 0 (none) to 3 (severe).
* Analgesic consumption. Analgesic consumption will be measured by recording the analgesics administered to the study subjects.
* Clinical recovery. Postoperative parameters will be recorded including time to clear fluid intake, voiding, and discharge from the hospital. The incidence of post-operative complications, such as post-operative nausea and vomiting and post-operative infections, will be noted as well.
* Global health questionnaire (GHQ). The GHQ is used to assess post-operative recovery; items include sleep, strength and energy, self-assistance and movement. The subjects rate every item on a six point Likert scale. The individual ratings are summed for a total recovery score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose health status is American Society of Anesthesiologists (ASA) physical status I to II, aged 10-21, with idiopathic scoliosis or congenital deformity of the chest wall, who are undergoing Nuss procedure/scoliosis repair at the Nationwide Children's hospital.
2. Parents/Guardian willing and able to authorize informed consent
3. Patients willing and able to authorize assent

Exclusion Criteria:

1. ASA classification III, IV (children with a chronic or severe disease).
2. Children with neuromuscular disorders
3. Children with developmental delay
4. Patients with preexisting mental illness

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pre-operative anxiety | Day of surgery, just prior to the procedure
  The STAI, completed by the patient to chart their own anxiety level, is a 40-item self-report measure that contains 20 items measuring state anxiety and 20 items measuring trait anxiety. Subjects are asked to respond on a 4-point Likert scale. Total scores for state and trait portions separately range from 20 to 80, with higher scores denoting higher levels of anxiety.
Post-operative pain | 24 hours post-op
  Total opiate consumption in the first 24 hours will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States